CLINICAL TRIAL: NCT06694805
Title: A Phase 3b, Open Label, Randomized, standard-of Care Control Arm, Multicenter, Superiority Study Evaluating the Efficacy, Safety, and Tolerability of Injectable CAB LA + RPV LA in Viremic Participants Living With HIV-1 (CROWN)
Brief Title: A Study to Evaluate the Effectiveness of Long-acting (LA) Cabotegravir (CAB) + Rilpivirine (RPV) LA When Given to Participants With Detectable HIV-1
Acronym: CROWN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221611; 2024-515070-28-00 (Other: EU CT)
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: HIV Infection; Cabotegravir; Rilpivirine; Long-acting; Efficacy; Safety; Durability
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CAB LA + RPV LA Group (Experimental): Participants receive initial injections at Day 1 and Month 1, followed by maintenance injections every 2 months for up to 24 months.
  Interventions: Drug: CAB LA + RPV LA
- Oral ART Control Group (Active Comparator): Participants continue to take their current oral ART for 6 months, including a final dose at their first injection visit.
  Interventions: Drug: Oral ART

INTERVENTIONS:
Drug: CAB LA + RPV LA — Intramuscular injection administered monthly for first 2 initiation doses then every 2 months.
  Arms: CAB LA + RPV LA Group
Drug: Oral ART — Oral medication provided to participants by the site/their regular healthcare professional (HCP) as part of their standard of care (SOC) treatment.
  Arms: Oral ART Control Group

SUMMARY:
This study will assess how effective, safe, and long-lasting a long-acting antiretroviral therapy (ART) using CAB LA + RPV LA is for people with HIV who still have detectable virus levels despite being on oral ART. The study will also consider feedback from patients on their experience with this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age

  1. Aged >=12 years and >=35 kg (at the time of obtaining informed consent).
* Type of Participant and Disease Characteristics 2.HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA VL.

  3.Plasma HIV-1 RNA >1 000 c/mL and greater than (<) 100 000 c/mL at Screening. 4.Evidence of insufficient virologic response to participant's current oral ART regimen within 18 months prior to study entry according to at least 1 of the following criteria: i.<1 log10 decrease in HIV-1 RNA or HIV-1 RNA >200 c/mL at 2 time points at least 4 weeks apart in individuals who have been prescribed oral ART for at least 3 consecutive months.

ii. Documented lapse in current oral ART regimen usage expected to result in HIV-1 viremia (defined as at least a 30-day consecutive period of non-use of oral ART) iii. Documented need for change from oral ART regimen that investigator attributes as primary reason for insufficient virologic response (e.g., safety findings and/or limited tolerability, clinically relevant DDIs).

Currently being treated with an oral ART regimen specific regimen to be recorded at Screening, and willing to continue taking that regimen until approximately 1 week after the Month 6 visit.

* Pregnancy, Sex and Contraceptive/Barrier Requirements 5. Person of childbearing potential (POCBP) must have a negative serum or urine pregnancy test at screening and on Day 1.
* Informed Consent/Assent 6.Informed consent/Assent must be provided as follows:

  1. Adult participants (>=18 years old) must be capable of giving signed informed consent as described in the full study protocol, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and stated in the full study protocol.
  2. For adolescent participants (12 to <18 years of age at screening), the parent(s) or legal guardian must be capable of giving signed informed consent.

Exclusion Criteria:

• Medical Conditions

1. HIV-1 Subtype A6, if known from historical result.
2. Participants who are pregnant, breast/chest feeding or plan to become pregnant or breast/chest feed during the study.
3. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones).
4. Individuals with both HIV and Hepatitis B virus (HBV) will be excluded from participating in studies where they would not be able to receive appropriate therapy for their HBV co-infection and therefore may be at risk of hepatitis B flare. Exclusion will be determined by evidence of HBV infection based on the results of testing at Screening for HBsAg, HBcAb, HBsAb and HBV.
5. History of liver cirrhosis with or without hepatitis viral co-infection.
6. Participants with severe hepatic impairment (Class C) as determined by Child-Pugh classification.
7. Participants with HCV co-infection will be excluded entry into this study if they are currently receiving anti-HCV therapy at baseline (Day 1).
8. Participants determined by the investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder.
9. History of sensitivity to any of the study medications or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
10. Participants who in the investigator's judgment, pose a significant suicidality risk. Participant's history of suicidal behaviour and/or suicidal ideation should be considered when evaluating for suicide risk.
11. Any pre-existing physical or mental condition which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.

    • Prior/Concomitant Therapy
12. Any previous use of CAB.
13. Current or anticipated need for chronic anti-coagulants.
14. Use of concomitant medications which are associated with Torsades de Pointes (TdP).
15. Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
16. Treatment with any of the following agents within 28 days of Screening:

    1. radiation therapy;
    2. cytotoxic chemotherapeutic agents;
    3. tuberculosis therapy with the exception of isoniazid;
    4. anti-coagulation agents, with the exception of the use of low dose acetylsalicylic acid (<=325mg);
    5. immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons.
17. Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigational medicinal product (IP).
18. Participants receiving any protocol-prohibited medication and who are unwilling or unable to switch to an alternate medication.

    • Prior/Concurrent Clinical Study Experience
19. Participant is currently participating in, or anticipates being selected for, any other interventional study.

    • Diagnostic assessments
20. Any evidence of viral drug resistance based on the presence of any major RAM to INSTIs or NNRTIs in the Screening result; or, if known, in any historical resistance test result.
21. Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's participation in the study of an investigational compound.
22. Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 lipid abnormalities. A single repeat test is allowed during the Screening period to verify a result.
23. ALT >=5 times ULN or ALT >=3×ULN and bilirubin >=1.5×ULN (with >35% direct bilirubin).
24. eGFR of <30 mL/min/1.73 m2 via refitted, race-neutral CKD-EPIcr_R method (adult participants) or <50 mL/min/1.73 m2 using the Bedside Schwartz equation (adolescent participants).
25. Hemoglobin <9.0 g/dL.
26. Corrected QT interval (QTc >450 msec or QTc >480 msec for participants with bundle branch block, calculated using ECGs performed in triplicate).

    • Other exclusions
27. Unwilling to receive injections, or unable to receive gluteal injections.
28. The participant has gluteal implants or prosthesis; or a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reaction (ISRs).
29. Evidence of alcohol or substance use disorder within the previous 12 months, using standard methods for their site, that would interfere with the participant's safety.
30. Adolescents who are wards of the state or government. To assess any potential impact on participant eligibility with regard to safety, the investigator must refer to the Investigator's brochure (IB) and supplements, approved product labels, and/or local prescribing information for detailed information regarding warnings, precautions, contraindications, AEs, drug interactions, and other significant data pertaining to the study drugs.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2028-06-19 (Estimated)

PRIMARY OUTCOMES:
Number of participants with virologic suppression after the CAB LA + RPV LA treatment compared to oral ART | At Month 6
  A virologic suppression is defined by HIV-1 RNA less than (<) 50 copies (c)/mL.

SECONDARY OUTCOMES:
Time to virologic suppression | From Baseline (Day 1) up to Month 6
Time to treatment related discontinuation (=Failure) (TRDF) | From Baseline (Day 1) up to Month 6
  TRDF can be caused by a confirmed virologic failure or a drug-related adverse event (AE), intolerability of injections, protocol defined stopping criteria or lack of efficacy.
Number of participants with confirmed protocol-defined virologic failure (VF) | From Baseline (Day 1) up to Month 6
  VF is defined as: confirmed plasma HIV-1 RNA levels greater than or equal to (>=) 400 c/mL on or after Month 4; confirmed rebound in plasma HIV-1 RNA levels to >=400 c/mL after prior confirmed suppression to <400 c/mL; confirmed plasma HIV-1 RNA levels greater than (>) 1 log10 c/mL above the nadir value where nadir is >=400 c/mL; decrease in plasma HIV-1 RNA of <1 log10 c/mL by Month 1, with subsequent. confirmation, and resistance emergence to ARVs (unless plasma HIV-1 RNA is. <400 c/mL).
Number of participants with treatment-emergent resistance-associated mutations (RAMs) | From Baseline (Day 1) up to Month 6
Number of participants with treatment-emergent RAMs | Up to Month 12 and Month 24
Number of participants with serious adverse events (SAEs) | Up to Month 6, Month 12, and Month 24
  A SAE is defined as any untoward medical occurrence that, at any dose, meets one or. more of the following criteria: results in death, is life threatening, requires inpatient hospitalization (or prolongation of existing hospitalization), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, abnormal pregnancy outcomes and other significant medical events deemed so by the investigator.
Number of deaths | Up to Month 6, Month 12, and Month 24
Number of participants with Grade 2 to 5 drug-related adverse events (AEs) | Up to Month 6, Month 12, and Month 24
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not. considered related to the study intervention. Every AE is graded according to the DAIDS toxicity scales. Grade 2 = moderate symptoms, Grade 3 = severe symptoms, Grade 4 = Potentially life-threatening. symptoms and Grade 5 = death.
Number of AEs leading to discontinuation | Up to Month 6, Month 12, and Month 24

CONTACTS AND LOCATIONS:
Locations (62):
- United States (33):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Hawthorne, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (5):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Rosario
- GSK Investigational Site, Antwerp, Belgium
- GSK Investigational Site, Montreal, Quebec, Canada
- Germany (5):
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Düsseldorf
  - GSK Investigational Site, Frankfurt
- Italy (3):
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Roma
- GSK Investigational Site, Porto, Portugal
- GSK Investigational Site, San Juan, Puerto Rico
- Spain (12):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Sabadell Barcelona
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Vigo Pontevedra
  - GSK Investigational Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Study sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf